CLINICAL TRIAL: NCT02267278
Title: Evaluation of Ruxolitinib and Pracinostat Combination as a Therapy for Patients With Myelofibrosis
Brief Title: Ruxolitinib and Pracinostat Combination Therapy for Patients With Myelofibrosis (MF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0445; NCI-2015-00002 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Myeloproliferative Diseases
Keywords: Myeloproliferative Diseases; Myelofibrosis; MF; Primary or post essential thrombocythemia/polycythemia vera; Ruxolitinib; Jakafi; INCB018424; INC424; Pracinostat; Questionnaire; Survey
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — ruxolitinib; SB939 compound; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib + Pracinostat (Experimental): Ruxolitinib starting dose 15 mg orally twice/day in 28-day cycle (dose assigned based on platelet count, if low platelet count gradual up-titration from a starting dose of 5 mg) - given alone for first 3 months, then Pracinostat added at starting dose 60 mg orally once/day for 3 alternating days every 3 weeks starting Day 1 of Cycle 4.
  Dose of Ruxolitinib may be increased or decreased prior to initiation of Pracinostat. Quality of Life Questionnaire.
  Interventions: Drug: Ruxolitinib; Drug: Pracinostat; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib taken by mouth 2 times each day in a 28-day cycle. Patients receive Ruxolitinib alone for first 3 months, and then Pracinostat added. Starting dose of Ruxolitinib based on patients' platelet count. Dose of Ruxolitinib may be increased or decreased at discretion of treating physician prior to initiation of Pracinostat.
  Other Names: Jakafi; INCB018424; INC424
Drug: Pracinostat — Starting dose of Pracinostat 60 mg by mouth 1 time each day for 3 alternating days every 3 weeks starting on Day 1 of Cycle 4.
Behavioral: Questionnaire — Questionnaire regarding quality of life completed at baseline, within 3 days before Day 1 of Cycles 1 - 6, and then every 3 cycles after that.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if pracinostat, when given in combination with ruxolitinib, can help to control myelofibrosis (MF). The safety of this drug combination will also be studied.

This is an investigational study. Pracinostat is not FDA-approved or commercially available. It is currently being used for research purposes only. Ruxolitinib is FDA-approved and commercially available to treat MF.

The study doctor can explain how the study drugs are designed to work.

Up to 25 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take ruxolitinib by mouth 2 times each day. You may take your dose of ruxolitinib with or without food.

You will also take pracinostat by mouth 1 time each day for 3 alternating days (for example Monday, Wednesday, Friday or Tuesday, Thursday, Saturday) every 3 weeks starting on Day 1 of Cycle 4. You will take your dose of pracinostat in the morning, about 30 minutes before or 2 hours after a meal. You should swallow your dose of pracinostat whole with a cup of water (about 8 ounces).

You will be given a study drug diary to write down when you take your dose of study drugs and if you miss or vomit any doses of study drug. You must bring the diary with you to the clinic on Day 1 of each cycle and at the end-of-treatment visit. You will also need to bring any leftover pills and any empty containers of the study drugs to the clinic when the study doctor tells you to do so.

Study Visits:

There are 28 days (4 weeks) in every study cycle. You will visit MD Anderson for regular study visits while participating in this study during Cycles 2-7, and then once every 3 cycles after that (Cycles 10, 13, 16, and so on).

Once during Cycles 2-7 and then once every 3 cycles after that (Cycles 10, 13, 16, and so on):

* You will have a physical exam.
* You will complete the questionnaire about your quality of life.

At your visits during Cycles 4, 5, and 6 and then once every 3 cycles starting with cycle 10 (cycles 10, 13, 16 and so on): You will have an EKG to check your heart function.

At your visits during Cycles 4, 5, and 7 and then every 3 cycles after that (Cycles 10, 13, 16, and so on) blood (about 1-2 teaspoons) will be drawn for cytokine testing.

At your visits during Cycles 7 and 13, and then every 6 cycles after that (Cycles 19, 25, 31, and so on), if the doctor thinks it is needed, you will have a bone marrow biopsy to check the status of the disease and for cytogenetic and genetic testing.

Every 2 weeks during the first 6 cycles and then about every 3 cycles after that, blood (about 2-3 tablespoons) will be drawn for routine tests. In between the mandatory visits to MD Anderson, you may choose to have these blood draws performed at a local lab or clinic closer to your home. The results will be sent to the study doctor.

Length of Treatment:

You may continue taking the study drugs for up to 4 years. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up.

Follow-Up:

About 30 days after your last dose of study drugs, if you are not receiving another treatment for MF, you will be called by the study doctor or a member of the study staff and asked about any side effects you may be having. This call should last about 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MF (either primary or post essential thrombocythemia/polycythemia vera) requiring therapy, including those previously treated and relapsed or refractory, or if newly diagnosed, with intermediate-1 or -2 or high risk according to International Prognostic Scoring System (IPSS).
2. Palpable splenomegaly of more than or equal to 5 cm below left costal margin on physical exam
3. Understanding and voluntary signing an Institutional Review Board (IRB)-approved informed consent form.
4. Age equal to or more than 18 years at the time of signing the informed consent.
5. Disease-free of other malignancies.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
7. Negative pregnancy test in females of childbearing potential (FCBP). Male patients with female partners of child-bearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 30 days following last dose. Acceptable forms of contraception include 1 highly effective method such as an intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation, or partner's vasectomy and at least 1 additional approved barrier method such as a latex condom, diaphragm, or cervical cap. Female patients of childbearing potential must not be breast-feeding or planning to breast feed and must have a negative pregnancy test ≤7 days before first study treatment.
8. QTcF interval equal to or less than 470 msec
9. Normal serum potassium magnesium levels
10. Adequate organ function as demonstrated by the following: Direct bilirubin equal to or less than 2.0 mg/dL, Serum creatinine equal to or less than 2.0 mg/dL., Alanine transaminase (SGPT) equal to or less than 3 x upper limit of normal (unless considered to be related to MF or patient has known history of Gilberts)
11. Platelets >/= 50000/uL
12. Absolute Neutrophil count (ANC) >/= 1000/uL

Exclusion Criteria:

1. Prior therapy with a JAK inhibitor (other than ruxolitinib for less than 3 months duration and currently on it) or HDACi. Patients that are currently on ruxolitinib for less than 3 months of therapy are eligible.
2. Use of any other standard or experimental therapy within 14 days of starting study therapy.
3. Lack of recovery from all toxicity from previous therapy to grade 1 or baseline.
4. Suspected pregnancy, pregnant or lactating females.
5. Any condition, including the presence of laboratory abnormalities, which in the opinion of the treating physician places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
6. Known positive for HIV or infectious hepatitis, type A, B or C.
7. Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
8. Cardiopulmonary function criteria: • Current unstable arrhythmia requiring treatment • History of symptomatic congestive heart failure • History of myocardial infarction within 6 months of enrollment • Current unstable angina • Family history of long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2015 to March 2017
Pre-assignment Details: Of the twenty-five participants who started the study, five never began pracinostat and are not considered evaluable for response.
Period: Overall Study
Arm/Group | Ruxolitinib + Pracinostat
Started | 25
Completed | 20
Not Completed | 5
Not completed — Proceeded to transplantation (allo-HCT) | 1
Not completed — transformation to acute leukemia (AML) | 1
Not completed — Developed new cancer diagnoses | 2
Not completed — prescribed prohibited medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib + Pracinostat
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 67 [56 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR), defined as a clinical improvement (CI), partial remission (PR), and complete remission (CR) according to the International Working Group (IWG) Criteria. Complete remission (CR): bone marrow blasts <5%, hemoglobin >/= 10, absolute neutrophil count (ANC) >/= 1000, platelets >/= 100, <2% immature myeloid cell, spleen and liver not palpable. Partial Response (PR): CR plus one or more of the following: ANC >/= 1000, decreased platelets by 50%, hemoglobin >/= 8.5 but < 10, <2% immature myeloid cells. Clinical improvement (CI): hemoglobin increase of 2g/dl, transfusion independence or reduction splenomegaly and/or hepatomegaly >/= 50%, >/=50% reduction in MPN-SAF TSS
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib + Pracinostat
Number analyzed (Participants) | 20
Participants | 16

2. Secondary Outcome: Toxicity of Combination of Ruxolitinib With Pracinostat
Description: Toxicity defined as Grade 3-4 clinically relevant non-hematologic toxicity or a serious adverse event that is at least possibly related to the study drug (Common Terminology Criteria for Adverse Events CTCAE version 4.0).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib + Pracinostat
Number analyzed (Participants) | 20
Participants | 1

ADVERSE EVENTS:
Time Frame: up to three years
Description: All 25 participants registered on this study were evaluable for adverse events.
Arm/Group | Ruxolitinib + Pracinostat
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib + Pracinostat (N=25)
Benign Mass Kidney (Renal and urinary disorders) | 1 (1)
Bronchial Infection (Infections and infestations) | 1 (2)
Chest Pain - Cardiac (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 2 (4)
Conduction disorder (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stent placement (Surgical and medical procedures) | 1 (1)
Total Aurilectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib + Pracinostat (N=25)
Abdominal pain (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 17 (17)
Elevated Liver Function Tests (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 8 (8)
Flatulence (Gastrointestinal disorders) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Shingles (Skin and subcutaneous tissue disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13)
Weight gain (Investigations) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT02267278/Prot_SAP_000.pdf